CLINICAL TRIAL: NCT01489761
Title: Percutaneous Treatment of Very LONG Native Coronary Lesions With Drug-Eluting Stent-VI: Everolimus-eluting Versus Zotarolimus-Eluting Stents
Brief Title: LONG-DES VI (Drug Eluting Stent for Long Lesions in Coronary Artery)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: Abbott (Industry); CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVRF2011-9
Record Dates: First submitted 2011-12-08; First posted 2011-12-12 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Coronary Artery Disease
Keywords: long lesions; drug eluting stents
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zotarolimus-eluting stent (Active Comparator): Resolute Integrity or Resolute Onyx stent
  Interventions: Device: percutaneous coronary intervention
- everolimus-eluting stent (Experimental): Xience Prime or Xience Xpedition or Xience Alpine stent
  Interventions: Device: percutaneous coronary intervention

INTERVENTIONS:
Device: percutaneous coronary intervention — drug eluting stent implantation
  Other Names: Resolute Integrity or Resolute Onyx stent; Xience Prime or Xience Xpedition or Xience Alpine stent

SUMMARY:
This is a multi-center, randomized, study to compare the efficacy of zotarolimus-eluting stent (Resolute Integrity or Resolute Onyx stent) or everolimus-eluting stent (Xience Prime or Xience Xpedition or Xience Alpine stent) for very long coronary lesions.

DETAILED DESCRIPTION:
Following angiography, patients with significant diameter stenosis > 50% and lesion length (> 50mm) requiring at least 2 multiple long-stent placement by visual estimation and eligible for LONG-DES VI trial inclusion and exclusion criteria will be randomized 1:1 to zotarolimus-eluting stent (Resolute Integrity or Resolute Onyx stent) or everolimus-eluting stent (Xience Prime or Xience Xpedition or Xience Alpine stent) by the stratified randomization method.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 20 years
* Significant native coronary artery stenosis (> 50% by visual estimate) with lesion length of more than 50mm, which requires at least 2 multiple long stent placement without intervening normal segment
* Patients with silent ischemia, stable or unstable angina pectoris, and Non-ST-elevation myocardial infarction (NSTEMI)
* The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site

Exclusion Criteria:

* Any contraindication to any of the following medications: aspirin, heparin, clopidogrel, stainless steel, contrast agents, zotarolimus, or everolimus
* An elective surgical procedure is planned that would necessitate interruption of antiplatelet drugs during the first 6 months post enrollment
* Acute ST-segment-elevation MI or cardiogenic shock
* Terminal illness with life expectancy < 1 year
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period
* In-stent restenosis at target vessel (either bare metal stent or drug-eluting stent segment) However, non-target vessel In-stent restenosis is permitted
* Patients with EF < 30%
* Serum creatinine level >=2.0mg/dL or dependence on dialysis
* Patients with left main stem stenosis (> 50% visual estimate)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
In-segment late luminal loss at 13 month follow-up | 13 month post stenting

SECONDARY OUTCOMES:
1. All Death | 12 month clinical follow-up
2. Cardiac death | 12 month clinical follow-up
3. Myocardial infarction (MI) | 12 month clinical follow-up
4. Composite of death or MI | 12 month clinical follow-up
5. Composite of cardiac death or MI | 12 month clinical follow-up
6. Target vessel revascularization (ischemia-driven and clinically-driven) | 12 month clinical follow-up
7. Target lesion revascularization (ischemia-driven and clinically-driven) | 12 month clinical follow-up
8. Target-vessel failure (death from any cause, myocardial infarction, and ischemic-driven target-vessel revascularization) | 12 month clinical follow-up
9. Stent thrombosis (ARC criteria) | 12 month clinical follow-up
10. In-stent late loss | 13 month angiographic follow-up
11. In-stent and in-segment restenosis | 13 month angiographic follow-up
12. Angiographic pattern of restenosis | 13 month angiographic follow-up
13. Volume of intimal hyperplasia | 13 month IVUS follow-up
  sub-study
14. Incidence of late stent malapposition | 13 month IVUS follow-up
  sub-study
15. Procedural success defined as achievement of a final diameter stenosis of <30% by QCA using any percutaneous method, without the occurrence of death, Q wave MI, or repeat revascularization of the target lesion during the hospital stay | 2-3 days post stenting

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (11):
- South Korea (11):
  - Gangwon National Univ. Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National university hospital, Daegu
  - The Catholic University of Korea, Daejeon ST. Mary's Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - National Health Insurance Service Ilsan Hospital, Ilsan
  - Korea University Guro Hospital, Seoul
  - Kyunghee University Medical Center, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - St.carollo Hospital, Suncheon
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.